CLINICAL TRIAL: NCT04279093
Title: Digital Assessment of Well-being in New Parents (DAWN-P)
Brief Title: Digital Assessment of Well-being in New Parents
Acronym: DAWN-P
Status: Completed | Type: Observational
Sponsor: Emily Eisner (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor-Investigator, Emily Eisner, Research Associate, Manchester Academic Health Science Centre
Organization: Manchester Academic Health Science Centre (Other)
Other Study IDs: 274007
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Postnatal Depression
Keywords: digital screening; mental health; smartphone app; postnatal depression; maternal mental health; paternal mental health
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant/postpartum women and their partners: The investigators aim to recruit 20 women in late pregnancy from the Antenatal Assessment Unit and the Antenatal Clinic at St Mary's Hospital. Their partners will be invited to participate where applicable.
  Inclusion and exclusion criteria for pregnant women are as follows:
  * Inclusion: after 36 weeks gestation, aged over 18 years and fluent in English, under the care of Manchester University NHS Foundation Trust
  * Exclusion: current stillbirth (women experiencing a stillbirth during the study will be withdrawn from the study), fetal abnormality, or multiple pregnancy
  Inclusion criteria for partners: male or female partners of a mum participating in the study, aged over 18 and fluent in English.
  Interventions: Other: No intervention, but participants will use a smartphone app daily to complete the EPDS

INTERVENTIONS:
Other: No intervention, but participants will use a smartphone app daily to complete the EPDS — No intervention, but participants will use a smartphone app daily (ClinTouch DAWN-P) to complete the Edinburgh Postnatal Depression Scale

SUMMARY:
The mental health of new parents around the time of the birth of their baby has been identified as a key priority in the NHS (National Health Service) Long Term plan. At present, there is no nationally implemented method for monitoring parents' mental health, although the use of the Edinburgh Postnatal Depression Scale (EPDS) has been recommended. This is a paper based questionnaire administered by health visitors in the postnatal period. For the purposes of this project, the investigators contacted health visitors in Manchester to find out how they use EPDS in practice. Currently, health visitors only use the questionnaire if they feel there is a need during visits, and the questionnaire is not kept (only the overall score). Since almost 20% of mums develop postnatal depression, more systematic and thorough screening is needed.

The investigators developed an app version of the EPDS which takes less than 2 minutes to complete on a smartphone. It is anticpated that this will be a more accessible and practical method of conducting this important assessment. This project is a feasibility study to find out whether an app would be a feasible, acceptable, valid and safe way to monitor perinatal mental health in women and their partners.

The investigators aim to recruit 20 women and their partners in late pregnancy (after 36 weeks gestation) and ask them to use the app. The app will prompt completion of the EPDS once per day until 6 weeks postnatally. Participants' responses on the app will be transferred to a secure server at the University of Manchester. Participants will be invited to complete a paper version of the EPDS at the beginning and end of the study to check validity. They will also be asked to complete a questionnaire measuring the acceptability of the app and to take part in a brief qualitative interview at the end of the study.

ELIGIBILITY:
The investigators aim to recruit 20 women in late pregnancy from the Antenatal Assessment Unit and the Antenatal Clinic at St Mary's Hospital, Manchester. Their partners will be invited to participate where applicable.

Inclusion criteria for pregnant women:

* after 36 weeks gestation
* aged over 18 years
* fluent in English
* under the care of Manchester University NHS Foundation Trust

Exclusion criteria for pregnant women:

* current stillbirth (women experiencing a stillbirth during the study will be withdrawn from the study)
* fetal abnormality
* multiple pregnancy

Inclusion criteria for partners:

* male or female partners of a mum participating in the study
* aged over 18
* fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators aim to recruit 20 women in late pregnancy from the Antenatal Assessment Unit and the Antenatal Clinic at St Mary's Hospital, Manchester. Their partners will be invited to participate where applicable.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Percentage of app based EPDS (Edinburgh Postnatal Depression Scale) assessments completed during the app-use phase | 36 weeks gestation until 6 weeks postpartum
  Percentage of app based EPDS (Edinburgh Postnatal Depression Scale) assessments completed during the app-use phase
Percentage of eligible individuals recruited to the study | Baseline
  Percentage of eligible individuals recruited to the study
Dropout rate - percentage of participants who consent to take part in the study dropping out during the app use phase | 36 weeks gestation until 6 weeks postpartum
  Percentage of participants who consent to take part in the study dropping out during the app use phase
Percentage of participants completing at least a third of app-based assessments | 36 weeks gestation until 6 weeks postpartum
  Percentage of participants completing at least a third of app-based assessments. The a priori "accept" criterion will be >33% data points completed
Percentage of participants completing at least half of app-based assessments | 36 weeks gestation until 6 weeks postpartum
  Percentage of participants completing at least half of app-based assessments. The a priori target criterion will be 50% of participants submitting at least 50% of app-based assessments.

SECONDARY OUTCOMES:
Transcripts from qualitative interviews with parents who have used the screening app regarding acceptability of the app | 6 weeks postpartum
  Transcripts from qualitative interviews with parents who have used the screening app regarding acceptability of the app
abridged Mobile App Rating Scale | 6 weeks postpartum
  abridged Mobile App Rating Scale score
Edinburgh Postnatal Depression Scale - app-based version | 36 weeks gestation until 6 weeks postpartum
  Edinburgh Postnatal Depression Scale - app-based version
Edinburgh Postnatal Depression Scale - paper version | 36-37 weeks gestation; 5-6 weeks postpartum
  Edinburgh Postnatal Depression Scale - paper version
Number of adverse events occurring during the app-use phase of the study | 36 weeks gestation until 6 weeks postpartum
  Number of adverse events occurring during the app-use phase of the study
Qualitative interview data on participants' experience of using the app. | 6 weeks postpartum
  Qualitative interview data on participants' experience of using the app.
Demographic questionnaire | Baseline (36 weeks pregnant)
  Demographic questionnaire asking standard questions about participants' demographic characteristics - e.g. age, gender, employment status.
BMI (from casenotes) | Baseline (36 weeks pregnant)
  BMI (from casenotes)
past psychiatric history as reported in casenotes (any history of major depression, previously prescribed psychiatric medication, previously referred for talking therapy) | Baseline (36 weeks pregnant)
  past psychiatric history as reported in casenotes (any history of major depression, previously prescribed psychiatric medication, previously referred for talking therapy)
Answers to mental health screening questions at booking appointment (NICE, 2014: section 1.5.4) | Baseline (36 weeks pregnant)
  Answers to mental health screening questions at booking appointment (NICE, 2014: section 1.5.4)
Details of current childbirth (mode of delivery, live/still birth, any major obstetric complications) | Baseline (36 weeks pregnant)
  Details of current childbirth (mode of delivery, live/still birth, any major obstetric complications)
parity (total number of pregnancies reaching viable gestational age) | Baseline (36 weeks pregnant)
  parity (total number of pregnancies reaching viable gestational age)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of data beyond the research team will be on a per request basis; only that data which can be fully anonymised data will be shared.Qualitative data or full demographics will not be shared due to potential identifiability.

REFERENCES:
- [Derived] Eisner E, Lewis S, Stockton-Powdrell C, Agass R, Whelan P, Tower C. Digital screening for postnatal depression: mixed methods proof-of-concept study. BMC Pregnancy Childbirth. 2022 May 23;22(1):429. doi: 10.1186/s12884-022-04756-2. PMID 35606731

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04279093/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04279093/ICF_001.pdf